CLINICAL TRIAL: NCT01452867
Title: Comparison of Ventilation With Bag-Valve-Mask, Laryngeal Tube S-D and Laryngeal Mask Airway Supreme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Bruneck (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Gruber Elisabeth, Dr. med univ., Krankenhaus Bruneck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLS VENT 2011/04
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Cardiopulmonary Arrest
Keywords: Airway; Bag-Valve -Mask- Ventilation; Laryngeal Mask - Ventilation; Laryngeal Tube - Ventilation
MeSH Terms: conditions — Heart Arrest | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bag-Mask-Ventilation (Active Comparator): Bag-Valve Mask-Ventilation in 50 patients in general anesthesia
  Interventions: Device: Bag-Valve-Mask-Ventilation (Ambu Facemask)
- Laryngeal Mask Ventilation (Active Comparator): Laryngeal Mask Ventilation in 50 patients in general anesthesia
  Interventions: Device: Laryngeal Mask (Laryngeal Mask Airway Supreme)
- Laryngeal Tube Ventilation (Active Comparator): Laryngeal Tube Ventilation in 50 patients in general anesthesia
  Interventions: Device: Laryngeal Tube (Laryngeal Tube LT-S-D (VBM))

INTERVENTIONS:
Device: Bag-Valve-Mask-Ventilation (Ambu Facemask) — Bag-Valve Mask-Ventilation
  Other Names: Ambu Facemask
  Arms: Bag-Mask-Ventilation
Device: Laryngeal Mask (Laryngeal Mask Airway Supreme) — Ventilation
  Other Names: Laryngeal Mask Airway Supreme
  Arms: Laryngeal Mask Ventilation
Device: Laryngeal Tube (Laryngeal Tube LT-S-D (VBM)) — Ventilation
  Other Names: Laryngeal Tube LT-S-D (VBM)
  Arms: Laryngeal Tube Ventilation

SUMMARY:
Inexperienced rescuers may encounter severe problems in an unconscious patient in opening and maintaining an upper airway patent. Gaining evidence which ventilation technique may be most efficient and safe is of utmost importance to potentially improve outcome during cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
During cardiopulmonary resuscitation (CPR) ventilation has to be efficient to provide oxygen to the body and safe to avoid potentially fatal regurgitation and aspiration pneumonia and excessive stomach inflation. Basically trained rescuers have severe problems to ventilate a patient during cardiopulmonary resuscitation. This study intends to compare three commonly employed ventilation techniques. First, the traditionally bag-valve mask ventilation is commonly taught during CPR course, despite recent evidence suggesting low efficiency rates. Second, the laryngeal mask and the laryngeal tube supraglottic airways have shown high efficiency and safety in previous studies in the hand of experienced clinicians. Until now it is unclear if basically trained rescuers are better in ventilation with bag valve mask ventilation or the supraglottic airway devices, the laryngeal mask and the laryngeal tube. The purpose of this study is to compare in anesthetised patients airway management and ventilation with bag-valve mask, laryngeal mask and laryngeal tube.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

  -> 18 years old
* elective surgery in general anesthesia

Exclusion Criteria:

* Patient not sober
* BMI > 35kg/m2
* Pathologies of cerebral spine or peripheral neurological deficit
* Hiatus hernia, history of gastric reflux
* Stomach or Esophagus -Operation in the medical history
* Acute respiratory infection or obstructive lung disease
* Non elective surgery
* facial deformity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Airway Management time until first effective Ventilation | 90 sec
  Effective Ventilation within 90 Seconds required

SECONDARY OUTCOMES:
Stomach inflation | 60 sec
  Stomach inflation during ventilation with mask, laryngeal tube an laryngeal mask

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenhaus Bruneck, Bruneck, Bolzano, Italy